CLINICAL TRIAL: NCT01308931
Title: The Effect of Tubal Ligation, Essure Placement, AND Levonorgestrel Intrauterine Device on Serum Anti-Mullerian Hormone Rates Over Time
Brief Title: The Effect of Birth Control Methods on Anti-Mullerian Hormone (AMH) Levels
Status: Withdrawn | Type: Observational
Sponsor: Valleywise Health (Other)
Collaborators: Fertility Centers of Arizona (Other); St. Joseph's Hospital and Medical Center, Phoenix (Other)
Responsible Party: Sponsor
Other Study IDs: 2010-012
Record Dates: First submitted 2011-03-02; First posted 2011-03-04 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Birth Control
Keywords: Contraception; IUD; Essure; Tubal ligation; Anti-Mullerian hormone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Tubal ligation: Patients who elect to have tubal ligation
- Essure: Group that elects to have Essure placement
- Levonorgestrel IUD: Patients that elect to have a levonorgestrel intra-uterine device placement

SUMMARY:
Anti-mullerian hormone (AMH) has been shown to be a reliable marker of ovarian reserve. In prior studies, tubal ligation has been shown to have an adverse effect on ovarian reserve. One theory postulated for this effect is that the ovarian circulation is disrupted by the procedure, leading to altered hormone production. In this prospective cohort study, the investigators plan to analyze the rates of AMH decline by comparing the following contraceptive methods: tubal ligation, Essure placement, and levonorgestrel intrauterine devices (IUDs).

DETAILED DESCRIPTION:
Anti-mullerian hormone (AMH) has been shown to be a reliable marker of ovarian reserve because levels demonstrate a consistent age-related decline and do not fluctuate throughout the menstrual cycle. In prior studies measuring markers other than AMH, tubal ligation has been shown to have an adverse effect on ovarian reserve.

The primary aim of this study will be to compare the rates of anti-mullerian hormone (AMH) decline following tubal ligation, Essure placement, and levonorgestrel IUDs, and then identifying any and all differences that these specific contraceptive methods have on the changes of AMH rates over time. The secondary aim will focus on analyzing the various types of tubal ligation methods (i.e. coagulation, ligation, clips, bands, etc.) to see if different techniques result in any difference in the rate of AMH decline. The hypothesis is that tubal ligation will result in an accelerated rate of AMH decline as compared to other long-term or permanent contraceptive methods.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Female
* Age 25-40
* Electing one of the following contraceptive methods: tubal ligation, Essure, levonorgestrel IUD
* Ability to understand study procedures and to comply with them for the entire length of the study
* Willingness to comply with follow-up visit requirements

Exclusion Criteria:

* Age <25 or >40 at initiation or completion of the study
* Prior oophorectomy or salpingectomy
* Prior surgery of the ovaries or fallopian tubes
* Prior ovarian, uterine, or fallopian tube cancers
* Prior ovarian, uterine, or fallopian tube radiation exceeding >200rads
* Prior platinum-based or alkalizing chemotherapy
* Current cancer (any form)
* Current pregnancy
* Allergy to any of the components of the selected devices (titanium, rubber, nickel, plastic, silicone)
* Current drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements
* Inability or unwillingness of a potential participant to give written informed consent
* Inability for the potential participant to consent for herself

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women seeking contraceptive methods seen at Maricopa Integrated Health System, Fertility Centers of Arizona, or St Joseph's Hospital & Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-01; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Serum anti-Mullerian hormone levels | 24 months
  1 blood draw prior to procedure; four more blood draws at 6-month intervals

CONTACTS AND LOCATIONS:
Overall Officials: Daniel F Rychlik, MD, Principal Investigator — Maricopa Integrated Health System/Fertility Centers of Arizona
Locations (3):
- United States (3):
  - Maricopa Integrated Health System, Phoenix, Arizona
  - St Joseph's Hospital & Medical Center, Phoenix, Arizona
  - Fertility Centers of Arizona, Scottsdale, Arizona

REFERENCES:
- [Result] van Rooij IA, Broekmans FJ, Scheffer GJ, Looman CW, Habbema JD, de Jong FH, Fauser BJ, Themmen AP, te Velde ER. Serum antimullerian hormone levels best reflect the reproductive decline with age in normal women with proven fertility: a longitudinal study. Fertil Steril. 2005 Apr;83(4):979-87. doi: 10.1016/j.fertnstert.2004.11.029. PMID 15820810
- [Result] Goynumer G, Kayabasoglu F, Aydogdu S, Wetherilt L. The effect of tubal sterilization through electrocoagulation on the ovarian reserve. Contraception. 2009 Jul;80(1):90-4. doi: 10.1016/j.contraception.2008.12.012. Epub 2009 Mar 6. PMID 19501222